CLINICAL TRIAL: NCT02486016
Title: Determination of Serum Fentanyl Levels After Using Reference and Generic Transdermal Fentanyl TDSs With and Without Standardized Heat Application in Healthy Human Volunteers
Brief Title: Transdermal Patch CVD 2000: The Effect of Heat on Fentanyl Release From Fentanyl TDSs in Healthy Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Audra Stinchcomb, Principal Investigator, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: HP-00059884
Record Dates: First submitted 2015-06-26; First posted 2015-06-30 (Estimated); Results first posted 2019-09-10 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Peer Review, Research
Keywords: Bioequivalence; Therapeutic Equivalency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Duragesic Reference Fentanyl TDS (Experimental): Each volunteer participates in two procedure days using the Duragesic reference (RLD) fentanyl TDS with heating applied for one hour at hour 11 and hour 18, respectively.
  Interventions: Drug: Duragesic reference fentanyl TDS
- Apotex Generic Fentanyl TDS (Active Comparator): Each volunteer participates in two procedure days using the Apotex generic fentanyl TDS with heating applied for one hour at hour 11 and hour 18, respectively.
  Interventions: Drug: Apotex generic fentanyl TDS
- Mylan Generic Fentanyl TDS (Active Comparator): Each volunteer participates in two procedure days using the Mylan generic fentanyl TDS with heating applied for one hour at hour 11 and hour 18, respectively.
  Interventions: Drug: Mylan generic fentanyl TDS

INTERVENTIONS:
Drug: Duragesic reference fentanyl TDS — 25 µg/hour
  Other Names: Brand name fentanyl TDS
  Arms: Duragesic Reference Fentanyl TDS
Drug: Apotex generic fentanyl TDS — 25 µg/hour
  Other Names: Generic fentanyl TDS
  Arms: Apotex Generic Fentanyl TDS
Drug: Mylan generic fentanyl TDS — 25 µg/hour
  Other Names: Generic fentanyl TDS
  Arms: Mylan Generic Fentanyl TDS

SUMMARY:
This is an Open-label, Non-Randomized, 3-way Crossover Bioequivalence Study to compare fentanyl release after heating of a brand name (Duragesic) and generic (Apotex and Mylan) fentanyl (transdermal delivery system)TDSs in healthy adults.

DETAILED DESCRIPTION:
This research study is intended to determine the effect of heat on FDA-approved fentanyl TDSs and whether the heat applied will result in more fentanyl being absorbed through the skin than without applying heat. This is important given that little is known about how the release of fentanyl is affected by heat, particularly for generic products. This study will use fentanyl TDSs (brand name and generic TDSs) that have been approved by the Food and Drug Administration (FDA) and are already prescribed to customers in the United States, and will not include any placebos.

ELIGIBILITY:
Inclusion Criteria:

* 1. Men or non-pregnant women of any ethnic background between the age of 18 and 45 years old.
* 2. Subjects must be non-smokers (must have refrained from the use of nicotine-containing substances, including tobacco products (e.g., cigarettes, cigars, chewing tobacco, gum, patch or electronic cigarettes) over the previous 2 months and are not currently using tobacco products.
* 3. Provide written informed consent before initiation of any study procedures.
* 4. Available for follow-up for the planned duration of the study.
* 5. Able to communicate well with the investigators.
* 6. Able to adhere to the study protocol schedule.
* 7. Subjects who are within their ideal body weight (BMI>17 and ≤ 28).
* 8. Demonstrate comprehension of the protocol procedures and knowledge of study by passing (>70% correct responses) a written examination containing 20 multiple choice and true false questions covering all aspects of the study including the purpose, procedures, risks and benefits.
* 9. Subjects deemed to be healthy as judged by the Medically Accountable Investigator (MAI) and determined by medical history, physical examination, and medication history.
* 10. Negative urine drug screening test.
* 11. Have a normal blood pressure (systolic: 90-140 mmHg; diastolic: 50-90 mmHg) and heart rate (55-100 bpm).
* 12. Have normal screening laboratories for WBC, Hgb, platelets, sodium, potassium, chloride, bicarbonate, BUN, creatinine, ALT, AST and total bilirubin.
* 13. Have normal screening laboratories for urine protein and urine glucose.
* 14. Female subjects must be of non-childbearing potential (as defined as surgically sterile [i.e. history of hysterectomy or tubal ligation] or postmenopausal for more than 1 year), or if of childbearing potential must be non-pregnant at the time of enrollment and on the morning of each procedure, and must agree to use hormonal or barrier birth control such as implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), sexual abstinence, or a vasectomized partner.
* 15. Agrees not to participate in another clinical study during the study period.
* 16. Agrees not to donate blood to a blood bank throughout participation in the study and for at least 3 months after last procedure day.
* 17. Have a normal ECG.

Exclusion Criteria:

* 1. Women who are pregnant, lactating, breast feeding or have a positive serum pregnancy test at enrollment or on the morning of any procedure day.
* 2. Smokers (current use or use over the previous 2 months of nicotine-containing substances, including tobacco products (e.g., cigarettes, cigars, chewing tobacco, gum, patch or electronic cigarettes).
* 3. Participation in any ongoing investigational drug trial or clinical drug trial.
* 4. Abnormal Vital signs, defined as:

  * Hypertension (systolic blood pressure >140 mm Hg or diastolic blood pressure >90 mm Hg) at rest on 2 separate days)
  * Heart rate <55 at rest on 2 separate days
  * Respiratory rate >20
* 5. Temperature > 38.0°C (100.4°F) or symptoms of an acute self-limited illness such as an upper respiratory infection or gastroenteritis within 7 days of application of the fentanyl TDS.
* 6. History of chronic obstructive pulmonary disease.
* 7. Active positive Hepatitis B, C, and HIV serologies.
* 8. Positive urine drug screening test.
* 9. Use of any prescription medication during the period 0 to 30 days or over-the counter medication (vitamin, herbal supplements and birth control medications not included) during the period 0 to 3 days before entry to the study.
* 10. Donation or loss of greater than one pint of blood within 60 days of entry to the study.
* 11. Any prior serious adverse reaction or hypersensitivity to fentanyl, naltrexone or naloxone or any of the inactive ingredients in the TDS (alcohol, ethylene vinyl acetate-copolymer membrane and hydroxyethyl cellulose, polyester, silicone adhesive, isopropyl myristate, octyldodecanol, polybutene, polyisobutene, dimethicone NF, or polyolefin).
* 12. Have a diagnosis of schizophrenia or other major psychiatric diagnosis or mental illness (e.g. major depression).
* 13. Received an experimental agent (vaccine, drug, biologic, device, blood product or medication) within 1 month before enrollment in this study or expects to receive an experimental agent during the study.
* 14. Any condition that would, in the opinion of the Medically Accountable Investigator (MAI), place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.
* 15. Inability to communicate or co-operate with the investigators.
* 16. History of consumption of alcohol within 24 hours prior to dose administration.
* 17. Within 72 hours prior to dosing, use of antihistamines or use of topical drugs at TDS site.
* 18. Subject has an obvious difference in skin color between arms or the presence of a skin condition, open sore, scar tissue, tattoo, or coloration that would interfere with placement of test articles, skin assessment, or reactions to drug.
* 19. Use of monoamine oxidase inhibitors 21 days prior to study.
* 20. Failure to pass opioid dependence challenge test on each procedure day before application of the fentanyl TDS. Each subject will be injected subcutaneously with naloxone HCl (0.8 mg injection) and will be observed for 45 minutes for signs and symptoms of opioid withdrawal.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-07-09 (Actual); Primary Completion 2017-08-08 (Actual); Study Completion 2017-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Audra Stinchcomb, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore Center for Vaccine Development, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: AAPS presented poster — https://www.aaps.org/search?executeSearch=true&SearchTerm=published+posters&l=1 — Shin SH, Yu M, Thomas S, Hammell DC, Ghosh, P, Raney SG, Hassan HH, Stinchcomb AL. Evaluation of level A in vitro/in vivo correlations (IVIVC) for nicotine and fentanyl transdermal delivery systems with transient heat exposure by using multiple approaches. Poster presentation at the 2017 AAPS Annual Meeting and Exposition; November 12-15, 2017; San Diego, CA

RESULTS

PARTICIPANT FLOW:
Groups:
- Fentanyl TDS: Each volunteer participates in six procedure days. 1) Apotex generic fentanyl TDS (25 µg/h) with heat applied at 11 h for one hour 2) Apotex generic fentanyl TDS (25 µg/h) with heat at 18 h for one hour 3) Duragesic fentanyl TDS (25 µg/h) with heat applied at 11 h for one hour 4) Duragesic fentanyl TDS (25 µg/h) with heat at 18 h for one hour 5) Mylan generic fentanyl TDS (25 µg/h) with heat applied at 11 h for one hour 6) Mylan generic fentanyl TDS (25 µg/h) with heat at 18 h for one hour
  Two week wash out period between each procedure day.
Period: Overall Study
Arm/Group | Fentanyl TDS
Started | 10 (Same 10 volunteers completed Apotex, Duragesic and Mylan arms of the study; crossover study.)
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Same 10 volunteers used for all arms of the study; crossover study. The 10 volunteers were their own baselines.
Groups:
- Fentanyl TDS: Each volunteer participates in six procedure days.
  1. Apotex generic fentanyl TDS (25 µg/h) with heat applied at 11 h for one hour
  2. Apotex generic fentanyl TDS (25 µg/h) with heat at 18 h for one hour
  3. Duragesic fentanyl TDS (25 µg/h) with heat applied at 11 h for one hour
  4. Duragesic fentanyl TDS (25 µg/h) with heat at 18 h for one hour
  5. Mylan generic fentanyl TDS (25 µg/h) with heat applied at 11 h for one hour
  6. Mylan generic fentanyl TDS (25 µg/h) with heat at 18 h for one hour
  Two week wash out period between each procedure day.
Arm/Group | Fentanyl TDS
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Partial Area Under the Curve (AUC) Attained With Early and Late Heat in Each of the Three Fentanyl TDSs (Reference and Generic)
Description: Partial area under the flux-time curve of fentanyl calculated from 11 to 14 h for Early Heat and 18 to 21 h for Late Heat study designs
  Blood samples obtained at 15 min prior to patch application [baseline], and at 1:00, 10:00, 10:55, 11:05, 11:15, 11:25, 11:35, 11:45, 12:00, 13:00, 14:00, 16:00, 17:00, 17:55, 18:05, 18:15, 18:25, 18:35, 18:45, 19:00, 20:00, 21:00, and 22:00 h post-patch application
Time Frame: six procedure days for each participant
Population: Partial area under the flux-time curve of fentanyl from 11 to 14 h for Early Heat and 18 to 21 h for Late Heat study designs. Each was corrected to account for different TDS sizes. Comparison was early heat to late heat differences.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Apotex Generic Fentanyl TDS | Duragesic Reference Fentanyl TDS | Mylan Generic Fentanyl TDS
Number analyzed (Participants) | 10 | 10 | 10
h*ng/mL
  Early Heat (11 h) | 2.2 (1.4) | 1.7 (1.4) | 2.1 (1.8)
  Late Heat (18 h) | 2.7 (1.4) | 2.4 (1.0) | 2.9 (1.5)

ADVERSE EVENTS:
Time Frame: Minimum 19 weeks; the period of time was dependent on how long it took the volunteer to complete six procedure days with a minimum of 2 weeks washout between procedure days.
Arm/Group | Apotex Generic Fentanyl TDS | Duragesic Reference Fentanyl TDS | Mylan Generic Fentanyl TDS
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10 | 10/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apotex Generic Fentanyl TDS (N=10) | Duragesic Reference Fentanyl TDS (N=10) | Mylan Generic Fentanyl TDS (N=10)
Bradycardia (Cardiac disorders) | 9 (11) | 8 (12) | 5 (8)
Decreased respiratory rate (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (7) | 6 (8)
Increased respiratory rate (Respiratory, thoracic and mediastinal disorders) | 9 (15) | 10 (15) | 7 (10)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Increased blood pressure (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (2)
Abdominal cramping (Gastrointestinal disorders) | 3 (4) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Stat Plan (2017-06-12): https://cdn.clinicaltrials.gov/large-docs/16/NCT02486016/Prot_SAP_000.pdf
  • Statistical Analysis Plan: Stat Plan (2017-06-12): https://cdn.clinicaltrials.gov/large-docs/16/NCT02486016/SAP_001.pdf